CLINICAL TRIAL: NCT01590706
Title: An Association Study of Characterizing Cognitive Decline and Functional Cardiac Senescence Profile Through the Association of Biomarkers and Clinical Outcomes in Healthy Middle Aged and Elderly Korean Volunteers
Brief Title: A Study of Characterizing Cognitive Decline and Functional Cardiac Senescence in Healthy Korean Volunteers
Status: Completed | Type: Observational
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Collaborators: Daejeon University (Other)
Responsible Party: Principal Investigator, Dal-Seok Oh, OMD, PhD, Senior Investigator, Korea Institute of Oriental Medicine
Other Study IDs: KC1101
Record Dates: First submitted 2012-05-01; First posted 2012-05-03 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Aging; Mild Cognitive Impairment; Angina Pectoris
Keywords: Genotype-Phenotype Association; Aged; Middle Aged; Mild Cognitive Impairment; Heart Rate Control; Biomarkers
MeSH Terms: conditions — Cognitive Dysfunction; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples for single nucleotide polymorphism, and for cardiac enzyme level detection
Oversight: Data Monitoring Committee: Yes

SUMMARY:
* Although aging process appears to be generally characterized, investigators have been paid much attention to the specific target molecules, which leads to discover the clinical markers of the senescence. The present study is to investigate the clinical and biological profile of cognitive decline and functional cardiac senescence in healthy middle aged and elderly Korean volunteers.
* This study was conducted as a cross-sectional, single-center, comparative clinical study.
* Each volunteer was given informed consent for checking cognition and cardiac function. Blood and urine samples were collected to analyze genome, proteome, and metabolome to assess cognition and cardiac function of its muscle enzymes.

DETAILED DESCRIPTION:
* The protocol of this study was developed as the first assessment of the three to four series of clinical research on senescence.
* This design of the study is a non-interventional, single-center, single-visit design for investigating the cognitive decline and cardiac function including heart muscle enzyme activity, which have been considered one of the key points in aging process.
* Volunteers visit the study site during the screening period, informed consent for study participation and blood draw are given respectively, then, the eligibilities are met, participants visit the study site just once within two weeks.
* The participants undergo the following five procedures for 2-3 hours; out-patient visit,

  1. additional demographic interview including covariate factors (depression status, marital status
  2. vital sign check
  3. the questionnaire for cognitive function
  4. blood draw for genomic, proteomic, and metabolomic analyses (10 milli Liter), urine collection (20 milli Liter)
  5. electrocardiogram (ECG), then they are discharged.
* Their safety follow-up is monitored in a week (± 1 day) by a phone-call from the study associates.
* To evaluate cognitive function, several cognitive batteries were used, 3MSE (Modified-Mini Mental State Examination), ADAS-cog (Alzheimer's Disease Assessment Scale-cognitive subscale); for cognitive biomarkers, Apolipoprotein E, Type-3 metabotropic glutamate receptors.
* To evaluate cardiac function including its enzyme activity: HRV (heart rate variability), CRP (c-reactive protein); Cardiac Troponin T.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects >= 45 and <= 80 years of age
* who understands the study procedures signs informed consent forms

Exclusion Criteria:

* who > 150 mmHg in systolic or < 95 mmHg in diastolic blood pressure
* who > 110 mg/dl in fast glucose level
* Smoking > 20 cigarettes/day
* Alcohol > 3 units/day (1 unit = pure alcohol 10 milli Liter)
* Caffeine > 5 cups of coffee or tea/day

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy middle aged (45-64 age) and elderly (over 65 age) person
Sampling Method: Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miyoung Lee, PhD, Study Director — Korea Institute of Oriental Medicine
Locations (1):
- Dunsan Oriental Hospital of Daejeon Univ., Daejeon, South Korea